CLINICAL TRIAL: NCT02133560
Title: Use of Mobile Technology for Intensive Training in Medication Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Sicklesoft Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052665
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Sickle Cell Disease; Thalassemia
Keywords: Sickle cell; Thalassemia; Adherence
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Videotape Recording; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medication Administration + Education (Other): Subjects will be asked to monitor their daily iron chelator administration by taking a video recording of preparing it and ingesting at least one sip during months 1-3 and completing the medication administration log during months 1-6. During months 1-6 subjects will meet with study staff and receive educational materials on a monthly basis. The data collected will be analyzed to describe patient adherence and comfort level with the process of daily recording of medication management.
  Interventions: Behavioral: Video recording; Behavioral: Medication Administration Log; Behavioral: Education

INTERVENTIONS:
Behavioral: Video recording — Subjects will be asked to monitor their daily iron chelator administration by taking a video recording of preparing it and ingesting at least one sip. The data collected will be analyzed to describe patient adherence and comfort level with the process of daily recording of medication management.
Behavioral: Medication Administration Log — Subjects will be asked to monitor their daily iron chelator administration by completing the medication administration log on a daily basis. The data collected will be analyzed to describe patient adherence and comfort level with the process of daily recording of medication management.
Behavioral: Education — During this first six months period a study staff member will see subjects at each scheduled clinic visit they attend for regular blood transfusion.
  Subjects will receive educational material and short quizzes related to sickle cell disease, thalassemia, iron overload, or iron chelation.

SUMMARY:
Purpose: Assess whether intensive training with education and daily remote monitoring with provider involvement has a lasting positive impact on adherence to medication management. The study will seek to enroll 25 subjects with sickle cell disease or thalassemia, and less than 100% compliance for taking iron chelators in the previous three month prior to participation in the study. Subjects will be asked to monitor their daily iron chelator administration by taking a video recording of preparing it and ingesting at least one sip. Subjects will also use a medication log to record daily administration of medication, and meet with study staff monthly for educational activities. The data collected will be analyzed to describe patient adherence and comfort level with the process of daily recording of medication management. Mean percent adherence in the pre-study periods and each of the study periods will be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sickle cell or thalassemia
* History of iron overload

Exclusion Criteria:

* None

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-05; Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Increase adherence to medication regimen | Baseline, 3 month, 6 month, 12 month
  Assess whether intensive training with education and daily remote monitoring with provider involvement has a lasting positive impact on adherence to medication management. Mean percent adherence in the pre-study periods and each of the study periods will be analyzed and compared. The ANOVA will be performed to compare adherence to medication administration during periods of intensive interactions, period prior to study enrollment, and period post training during regular care follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmish Shah, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States